CLINICAL TRIAL: NCT06788171
Title: A Phase II Trial of PULSAR (Personalized Ultrafractionated Stereotactic Adaptive Radiotherapy) Combined With PD-1 Ab and Chemotherapy Plus Bevacizumab for Colorectal Cancer Liver Metastasis
Brief Title: PULSAR Combined With PD-1 Ab and Chemotherapy Plus Bev. for CRLM
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LIVERT
Record Dates: First submitted 2025-01-14; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Colorectal Cancer Liver Metastasis
MeSH Terms: interventions — Bevacizumab; Capecitabine; Oxaliplatin; sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PULSAR combined with PD-1 Ab and Bevacizumab plus Chemotherapy (Experimental): Interventions:
  1. Radiation: PULSAR(Personalized Ultrafractionated Stereotactic Adaptive Radiotherapy)
  2. Drug: Bevacizumab
  3. Drug: Capecitabine
  4. Drug: Oxaliplatin
  5. Drug: Sintilimab
  Interventions: Radiation: Personalized Ultrafractionated Stereotactic Adaptive Radiotherapy; Drug: Bevacizumab; Drug: Capecitabine; Drug: Oxaliplatin; Drug: Sintilimab

INTERVENTIONS:
Radiation: Personalized Ultrafractionated Stereotactic Adaptive Radiotherapy — PULSAR (SBRT): A targeted radiation therapy delivering 5-10 Gy/fraction every 3 weeks (q3w) to the gross tumor volume (GTV), for 3 times.
Drug: Bevacizumab — Bevacizumab: 5mg/kg, d1, q3w, 6 cycles.
Drug: Capecitabine — Capecitabine: 1000mg/m2, d1-14, bid, q3w, 6 cycles.
Drug: Oxaliplatin — Oxaliplatin: 130mg/m2, d1, q3w, 6 cycles.
Drug: Sintilimab — Sintilimab: 200mg, d1, q3w, 6 cycles.

SUMMARY:
To explore Progression-Free-Survival(FPS) of PULSAR(personalized ultrafractionated stereotactic adaptive radiotherapy) combined with PD-1 Ab and Chemotherapy plus Bevacizumabfor CRLM

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years, any gender.
2. Pathologically confirmed colorectal cancer with liver metastases (stage M1).
3. Karnofsky Performance Status ≥70.
4. Adequate organ function, no contraindications to radiotherapy, or immunotherapy.
5. Microsatellite/mismatch repair status MSS/pMMR.
6. No prior chemotherapy or any other anti-tumor treatment before inclusion.
7. No prior immunotherapy.
8. Ability to comply with the study protocol during the study period.
9. Signed written informed consent.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Pathological diagnosis of signet ring cell carcinoma.
3. History of other malignancies within the past 5 years, except cured skin cancer and cervical carcinoma in situ.
4. Uncontrolled epilepsy, central nervous system disorders, or history of psychiatric disorders that, in the opinion of the investigator, may interfere with signing the informed consent form or affect patient compliance with oral medication.
5. Clinically significant (i.e., active) cardiac disease, such as symptomatic coronary artery disease, New York Heart Association (NYHA) Class II or greater congestive heart failure, or significant arrhythmias requiring drug intervention (see Appendix 12), or history of myocardial infarction within the past 12 months.
6. Organ transplant recipients requiring immunosuppressive therapy and long-term steroid users.
7. Patients with autoimmune diseases.
8. Severe uncontrolled recurrent infections or other severe uncontrolled comorbidities.
9. Subjects with baseline hematological and biochemical parameters not meeting the following criteria: hemoglobin ≥90g/L; absolute neutrophil count (ANC) .≥1.5×10^9/L; platelets ≥100×10^9/L; ALT, AST ≤2.5 times the upper limit of normal; ALP ≤2.5 times the upper limit of normal; serum total bilirubin <1.5 times the upper limit of normal; serum creatinine <1 times the upper limit of normal; serum albumin ≥30g/L.
10. Known deficiency of dihydropyrimidine dehydrogenase (DPD).
11. Allergy to any investigational drug components.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free-Survival | From enrollment to 36 month

SECONDARY OUTCOMES:
Adverse Reactions | From enrollment to 36 month
Overall Survival (OS) | From enrollment to 36 month
Objective Response Rate (ORR) | From enrollment to 36 month

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Cancer Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No